CLINICAL TRIAL: NCT04815460
Title: Aerobic Interval and Moderate Continuous Exercise Training on Ventricular Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Chang Gung University (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 104-9615A3
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Healthy; High Intensity Interval Training; Exercise Training
Keywords: Stress echocardiography; Hypoxia test; Speckle-tracking echocardiography; High Intensity Interval Training
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity-interval training (HIIT) (Experimental): Subjects performed HIIT (3-min intervals at 40% and 80%VO2peak) on a bicycle ergometer for 30 min/day, 5 days/week for 6 weeks.
  Interventions: Behavioral: High intensity-interval training (HIIT)
- Ｍoderate intensity-continuous (MCT) (Experimental): Subjects performed MICT (sustained 60%VO 2max) on a bicycle ergometer for 30 min/day, 5 days/week for 6 weeks.
  Interventions: Behavioral: Moderate intensity-continuous (MICT)
- Control group (No Intervention): Without any exercise training

INTERVENTIONS:
Behavioral: High intensity-interval training (HIIT) — Subjects performed HIIT (3-min intervals at 40% and 80%VO2peak) on a bicycle ergometer for 30 min/day, 5 days/week for 6 weeks.
  Arms: High intensity-interval training (HIIT)
Behavioral: Moderate intensity-continuous (MICT) — Subjects performed MICT (sustained 60%VO 2max) on a bicycle ergometer for 30 min/day, 5 days/week for 6 weeks.
  Arms: Ｍoderate intensity-continuous (MCT)

SUMMARY:
Hypoxic exposure increases right ventricular (RV) afterload by triggering pulmonary hypertension, with consequent effects on the structure and function of the RV. Improved myocardial contractility is a critical circulatory adaptation to exercise training. However, the types of exercise that enhance right cardiac mechanics during hypoxic stress have not yet been identified. This study investigated how high-intensity interval training (HIIT) and moderate-intensity continuous training (MICT) influence right cardiac mechanics during hypoxic exercise (HE).

DETAILED DESCRIPTION:
Hypoxic exposure increases right ventricular (RV) afterload by triggering pulmonary hypertension, with consequent effects on the structure and function of the RV. Improved myocardial contractility is a critical circulatory adaptation to exercise training. However, the types of exercise that enhance right cardiac mechanics during hypoxic stress have not yet been identified. This study investigated how high-intensity interval training (HIIT) and moderate-intensity continuous training (MICT) influence right cardiac mechanics during hypoxic exercise (HE).

The young and healthy sedentary males were randomly selected to engage in either HIIT (3-min intervals at 40% and 80% of VO2 oxygen uptake reserve) or MICT (sustained 60% of VO2 oxygen uptake reserve) for 30 min/day and 5 days/week for 6 weeks or were included in a control group (CTL) that did not engage in any exercise. Right cardiac mechanics during semiupright bicycle exercise tests under hypoxic conditions (i.e., 50 watts under 12% FiO2 for 3 min) were measured using two-dimensional speckle-tracking echocardiography. The primary outcome was the change in right cardiac mechanics during semiupright bicycle exercise under hypoxic conditions (i.e., 50 watts under 12% FiO2 for 3 min) as measured by two-dimensional speckle tracking echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Having a sedentary lifestyle (without regular exercise, exercise frequency ≤ once weekly, duration < 20 min).

Exclusion Criteria:

* Exposed to high altitudes (> 3000 m) for at least 1 year.
* Smoker
* Taking medications or vitamins
* Having any cardiopulmonary/hematological risk.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
The changes of right cardiac mechanics during hypoxia stress echocardiography: Strain | 8 weeks
  1. Hypoxia stress echocardiography was collected under hypoxic conditions (12% FiO2) and used two-dimensional Speckle-tracking echocardiography.
  2. The resting images were acquired after the subject was placed in the aforementioned position for 10 min.
  3. The exercise images were conducted using semirecumbent cycling with a 50-Watt resistance for 3 min and acquired at the third minute of cycling to ensure that subjects had reached a steady-state HR (i.e., HR changes <10 bpm within 10 s and <110-120 bpm).
  4. A modified apical four-chamber view was used to assess 2D-STE longitudinal and radial parameters of the RV and RA.
  5. The RV strain was calculated using the average peak segmental values displayed by the software using a 6-segment model.
The changes of right cardiac mechanics during hypoxia stress echocardiography: Strain rate | 8 weeks
  1. Hypoxia stress echocardiography was collected under hypoxic conditions (12% FiO2) and used two-dimensional Speckle-tracking echocardiography.
  2. The resting images were acquired after the subject was placed in the aforementioned position for 10 min.
  3. The exercise images were conducted using semirecumbent cycling with a 50-Watt resistance for 3 min and acquired at the third minute of cycling to ensure that subjects had reached a steady-state HR (i.e., HR changes <10 bpm within 10 s and <110-120 bpm).
  4. A modified apical four-chamber view was used to assess 2D-STE longitudinal and radial parameters of the RV and RA.
  5. The RV strain rate was calculated using the average peak segmental values displayed by the software using a 6-segment model.

SECONDARY OUTCOMES:
Cardiopulmonary fitness | 8 weeks
  To assess cardiopulmonary fitness, cardiopulmonary exercise test (CPET) on a cycle ergometer was performed 4 days before and after the intervention. All subjects underwent exercise with a mask to measured oxygen consumption (VO2) breath by breath using a computer-based system (Master Screen CPX, Cardinal-health Germany).
The cavity diameters of RV | 8 weeks
  RV basal cavity diameter (RVD1), mid-cavity diameter (RVD2), and RV longitudinal diameter (RVD3), at end-diastole and end-systole, were evaluated in the modified apical four-chamber view.
Pulmonary vascular resistance (PVR) | 8 weeks
  Pulmonary vascular resistance (PVR) was calculated using the formula PVR = ([tricuspid regurgitation velocity/RVOT VTI] × 10 + 0.16)
  1. Tricuspid regurgitation velocity: Doppler imaging was used to measure peak tricuspid regurgitation velocities in systolic phase.
  2. The RV outflow tract (RVOT): obtained from a parasternal short-axis base view modified apical four-chamber view, and the flow immediately proximal to the pulmonary artery valve during systole was detected to calculate both maximal velocity and pulsed-wave blood velocity time integral (VTI)
RV diastolic function | 8 weeks
  Doppler imaging was used to measure peak tricuspid annular (E') and flow velocities (E) in early diastole.
Tricuspid annular plane systolic excursion (TAPSE) | 8 weeks
  Tricuspid annular plane systolic excursion (TAPSE) measures the longitudinal excursion of the tricuspid annulus in one dimension, which was measured by M-mode.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Shyan Wang, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Z, Chesler NC. Pulmonary vascular mechanics: important contributors to the increased right ventricular afterload of pulmonary hypertension. Exp Physiol. 2013 Aug;98(8):1267-73. doi: 10.1113/expphysiol.2012.069096. Epub 2013 May 10. PMID 23666792
- [Background] Jaijee S, Quinlan M, Tokarczuk P, Clemence M, Howard LSGE, Gibbs JSR, O'Regan DP. Exercise cardiac MRI unmasks right ventricular dysfunction in acute hypoxia and chronic pulmonary arterial hypertension. Am J Physiol Heart Circ Physiol. 2018 Oct 1;315(4):H950-H957. doi: 10.1152/ajpheart.00146.2018. Epub 2018 May 18. PMID 29775415
- [Background] Huang YC, Tsai HH, Fu TC, Hsu CC, Wang JS. High-Intensity Interval Training Improves Left Ventricular Contractile Function. Med Sci Sports Exerc. 2019 Jul;51(7):1420-1428. doi: 10.1249/MSS.0000000000001931. PMID 30829901
- [Background] Naeije R, Badagliacca R. The overloaded right heart and ventricular interdependence. Cardiovasc Res. 2017 Oct 1;113(12):1474-1485. doi: 10.1093/cvr/cvx160. PMID 28957537
- [Background] Fu TC, Wang CH, Lin PS, Hsu CC, Cherng WJ, Huang SC, Liu MH, Chiang CL, Wang JS. Aerobic interval training improves oxygen uptake efficiency by enhancing cerebral and muscular hemodynamics in patients with heart failure. Int J Cardiol. 2013 Jul 15;167(1):41-50. doi: 10.1016/j.ijcard.2011.11.086. Epub 2011 Dec 22. PMID 22197120